CLINICAL TRIAL: NCT05423184
Title: The Effectıveness Of Structured Myofascial Chain Exercise Training After Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Mirsad ALKAN, Principal Investigator, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023
Record Dates: First submitted 2021-12-08; First posted 2022-06-21 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Anterior Cruciate Ligament Injuries; Anterior Cruciate Ligament Rupture; Anterior Cruciate Ligament Tear
Keywords: Tele-Health; Sports injuries; Anterior Cruciate Ligament; Reconstruction; Exercise; Physical Therapy And Rehabilitation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Athletic Injuries; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Prospective Randomize Controlled Study
Who Masked: Participant
Masking Description: Knowledge that which exercises are structured for research will keep from participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise Therapy For Lower Extremities (Active Comparator): Participants will treated exercises with focused on lower extremities especilly knee joint and muscles. Exercise program continue for 18 sessions with 3 times a week and 6 week duration. Exercises are; straight leg raise, assisted squat, lunge. All sessions supervised by a physiotherapist with synchron tele-rehabilitation.
  Interventions: Other: Exercise Therapy For Lower Extremities
- Exercise Therapy For Myofascial Chains (Experimental): Participants will treated exercises with focused on whole body especilly myofascial chains.
  Exercise program continue for 18 sessions with 3 times a week and 6 week duration. Exercises are; straight leg raise, assisted squat, lunge with upper extremities and whole body participation. All sessions supervised by a physiotherapist with synchron tele-rehabilitation.
  Interventions: Other: Exercise Therapy For Myofascial Chains
- Control Group (No Intervention): Participants will do any exercises. They will join only assessment sessions.

INTERVENTIONS:
Other: Exercise Therapy For Lower Extremities — Participants who have inclusion criterias after ACL reconstrontion pos-op 8. week will included this study. Certified Physiotherapist who have master of science degree and doctorate student will assessed them before and after treatment with face to face. Also exercise education will give face to face with same therapist. After that first sessions patients will progress their standardize exercises pragram with telerehabilition during 6 weeks and 18 sessions. This program includes four directions single leg raise with theraband, squat, lunge walk and static balance exercises. All sessions will be supervised with physiotherapist. End of study assessments will perform again with same therapist.
  Arms: Exercise Therapy For Lower Extremities
Other: Exercise Therapy For Myofascial Chains — Participants who have inclusion criterias after ACL reconstrontion pos-op 8. week will included this study. Certified Physiotherapist who have master of science degree and doctorate student will assessed them before and after treatment with face to face. Also exercise education will give face to face with same therapist. After that first sessions patients will progress their structered exercises pragram with telerehabilition during 6 weeks and 18 sessions. This program includes four directions single leg and arm raise with theraband, squat with arm participation using theraband, lunge walk with arm participation using theraband and static balance exercises with arm participation using theraband. All sessions will be supervised with physiotherapist. End of study assessments will perform again with same therapist.
  Arms: Exercise Therapy For Myofascial Chains

SUMMARY:
Anterior cruciate ligament reconstruction(ACLR) surgery accepts best choices which condicions are totaly ruptured ACL or partial ruputures when patients with high activity level. Rehabilitation after ACL is an indispensable element of treatment because ACL injury causes severe instability and early degenerative changes in the knee. Although there is no standard rehabilitation program after ACLR but the concept of "Functional Rehabilitation" is prefers nowadays which structred according to therapeutic goals, it is planned in three stages as early, mid-term and late-term. After the late-term goals are achieved safely and the individuals reach to needed criterias, the stage of returning to sports or activity is planned. Patients with an active life expectancy, the goal at the end of rehabilitation after ACLR is to return to activity or sports and to reach pre-injury performance. Most individuals fail to return to sports or activity after ACL due to long-term strength deficits, neuromuscular and biomechanical changes, knee instability, and early developing knee osteoarthritis. Addition to that; changes that affect both the knee joint and the whole body biomechanics occur even in individuals who successfully return to activity and sports after ACL. Although there are problems that affect the whole body by exceeding a single segment in rehabilitation after ACLR; there is no study using the myofascial chain exercises approach in the treatment of these problems. Hip, core or trunk stabilization exercises and neuromuscular trainings that include more than one body segment added to the ACLR program provides more positive effects on rehabilitation outcomes than regional applications. In this project, researches aim to investigate that the effectiveness of structured myofascial chain exercises training, which will be applied in the late period of rehabilitation after ACLR, on functionality, performance and participation.In project scope; After completing the early and mid-term rehabilitation after surgery, the volunteers who met the criteria for transition to late rehabilitation were divided into two groups; lower extremity exercise training will be given to the first group and myofascial chain exercise training will be given to the second group. The control group will consist of healthy volunteers. In addition to the control group; The operated and intact extremities of the volunteers in the experimental groups will be compared. The training session, in which preterm and postterm evaluations and the exercises are taught, will be carried out with the face-to-face method, and the ongoing exercise sessions will be carried out with the telerehabilitation method. Reasearch outcome measures will be evaluated with strength, flexibility, balance, endurance, activity performance against time measurements and self-assessment questionnaires. End of this project; important data will be obtained in the fight against the risks created by the deficits that continue after the ACLR. The deficits seen after ACL fails to individuals from returning to their pre-injury functional level; the desired success cannot be achieved in returning to work, returning to sports, and returning to activity. Due to this situation, which poses a global problem, even if there is a return to work or sports after injury, branch and job changes may be required and the desired level of performance cannot be achieved. In individuals who cannot return to activity, inactive life increases the risk of non-communicable chronic diseases as well as the increased risk of osteoarthritis. In case of success in the project, important information will be obtained in order to prevent both the quality of life and the cost of secondary health and social life problems associated with ACL injuries. The content of the program will be expanded to include other sports injuries by applying to follow-up projects for the registration of the method to be applied for the first time.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-45
* Being able to establish written and verbal communication in Turkish
* Post-Op rehabilitation after primary ACL surgery with Autograft in reconstruction, at 8 weeks, post op at 12 weeks at the latest.
* To have participated in an exercise-based rehabilitation program structured by a physiotherapist in the early and mid-term after surgery (a standardized program will not be applied in the early and mid-term, and participation in the study after rehabilitation is sufficient)
* Gaining full range of motion in the knee joint in the direction of extension, gaining full range of motion in the flexion direction with a maximum loss of 5 degrees
* BMI greater than 20 and less than 30
* No previous history of surgery involving the lower extremity
* To be able to perform a normal gait pattern without compensatory movements
* m.Quadriceps Femoris Muscle strength of at least 60% of the healthy side
* Having an IKDC score of 55 or higher
* To have sufficient technological device usage skills and fast internet infrastructure to use video communication technologies without any problems.
* Having a device that provides the necessary equipment for video calling
* Having 15 m2 of space to allow exercise in the living area

Exclusion Criteria:

* Using allograft in reconstruction
* History of any chronic systemic, rheumatological, neurological, vascular disease
* History of traumatic injury to intact extremities and trunk in the last 6 months
* Presence of pain complaints including spine and shoulder pain over 3 according to the Visual Analogue Scale
* Those who use anti-inflammatory drugs
* Presence of cognitive or psychological illness that will prevent cooperation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
IKDC (International Knee Documentation Committee) Subjective Knee Score change is being assessed. | Change from Baseline knee function at 6 week
  Self-Reported measure score was recorded with higher scores mean better outcomes.

SECONDARY OUTCOMES:
Quadriceps Femoris and Hamstring muscle strength change is being assessed. | Change from baseline knee strength at 6 week
  Isometric muscle testing with digital hand held dynamometer was performed for three times. Maximum value of musle strenght in lbs were recorded.
Flexibility change is being assessed. | Change from Baseline flexibility at 6 week
  Sit and Reach Test was performed for three times. Maximum value of reaching in cm were recorded.
Static balance change is being assessed. | Change from Baseline Balance at 6 week
  Modified with flat ground flamingo balance test were performed for three times. Minimum number of faults in a minute were recorded.
Dynamic balance change is being assessed. | Change from Baseline Balance at 6 week
  Y Balance Test were performed for three times. Maximum value of reaching in cm were recorded.
Performance change is being assessed. | Change from Baseline Performance at 6 week
  Repeated sitting and stepping moves in 30 seconds were performed for three times. Maximum number of moves were recorded.
Lysholm Knee Score change is being assessed. | Change from Baseline knee function at 6 week
  Self-Reported measure score was recorded with higher scores mean better outcomes.
Knee injury and Osteoarthritis Outcome Score | Change from Baseline knee function at 6 week
  Self-Reported measure score was recorded with higher scores mean better outcomes.
Tampa Kinesiophobia | Change from Baseline kinesiophobia function at 6 week
  Self-Reported measure score was recorded with lower scores mean better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No